CLINICAL TRIAL: NCT00568828
Title: Pilot Study to Evaluate the Changes of Macular Pigment Optical Density in Patients With Idiopathic Macular Teleangiectasia Following Supplementation of Lutein and Zeaxanthin
Brief Title: MPOD in Macular Teleangiectasia Following Supplementation of Lutein and Zeaxanthin
Acronym: MacTEL-Supp
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Lowy Medical Research Institute Limited (Other)
Responsible Party: Daniel Pauleikhoff MD, Dep. of Ophthalmology, St. Franziskus Hospital, Muenster, Germany
Other Study IDs: MacTEL Supplement
Record Dates: First submitted 2007-12-05; First posted 2007-12-06 (Estimated); Last update posted 2007-12-06 (Estimated); Status verified 2007-12

CONDITIONS: Macular Teleangiectasia; Macular Pigment
Keywords: Macular Teleangiectasia; Macular Pigment

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Earlier investigations have detected low levels of macular pigment (MP) in the center of the fovea and a halo of MP at a higher eccentricity in persons with type 2 idiopathic juxtafoveal teleangiectasia (MACTEL)[Helb H-M, Charbel Issa P, Pauleikhoff D, Scholl HPN, Holz FG, MacTel-Study Group. Macular Pigment Density and Distribution in Patients with Macular Telangiectasia. ARVO Annual Meeting 2006, Fort Lauderdale, 30.04.-5.05.2006. Program # 5701/B795]. To date it is not known whether the total MP is reduced in MACTEL or whether even more MP accumulates at higher eccenticities compared to healthy probands. With the suggested study we aim to

1. investigate Lutein and Zeaxanthin serum levels in MACTEL probands
2. investigate and quantify MP at the posterior pole of MACTEL probands
3. detect possible changes of MP concentration and distribution following supplementation with Lutein and Zeaxanthin

DETAILED DESCRIPTION:
Rationale for performing this study Earlier investigations have detected low levels of macular pigment (MP) in the center of the fovea and a halo of MP at a higher eccentricity in persons with type 2 idiopathic juxtafoveal teleangiectasia (MACTEL)[Helb H-M, Charbel Issa P, Pauleikhoff D, Scholl HPN, Holz FG, MacTel-Study Group. Macular Pigment Density and Distribution in Patients with Macular Telangiectasia. ARVO Annual Meeting 2006, Fort Lauderdale, 30.04.-5.05.2006. Program # 5701/B795]. To date it is not known whether the total MP is reduced in MACTEL or whether even more MP accumulates at higher eccenticities compared to healthy probands. With the suggested study we aim to

1. investigate Lutein and Zeaxanthin serum levels in MACTEL probands
2. investigate and quantify MP at the posterior pole of MACTEL probands
3. detect possible changes of MP concentration and distribution following supplementation with Lutein and Zeaxanthin

The suggested study During this study we plan to select at least 10 MACTEL probands with different patterns of MP distribution including

1. those with detectable accumulation of MP in the center and segmental reduction of MP temporally
2. those with nearly no central accumulation and and larger area of reduced MP temporally
3. those with no detectable accumulation of MP in the center and a halo of MP at a more eccentric location These probands will be supplemented with Lutein (L) and Zeaxanthin (Z) (12mg L and 1 mg Z, provided as esters, 120mg Vitamin C, 17.6 mg Vitamin E, 10mg Zink, 40µg Selen (Ocuvite Lutein™)) for a duration of nine months. During the supplementation and three months after stop of supplementation, probands will be investigated every three months including

1. ophthalmologic investigation, 2. fundus photography, 3. measurement of MP with a modified Heidelberg retina Angiograph employing two excitation wavelengths (514 and 488nm) 4. measurement of L and Z in serum.

Aim of the study

1. Investigation of changes of MP concentration and distribution following supplementation of L and Z in MACTEl probands
2. How do serum levels of L and Z change in these probands?

Visit:

V1 Screening & Start of supplementat V2 V3 V4 End of supplemenation V5 after stop of intake Months 0 3 6 9 12 general Informed consent X Medical history X in- and exclusion criteria X concommitant medication X X X X X Adverse events X X X X Pill count X X X Vital signs/ BMI X X Slitlamp investigation X X X X X Fundusphotography X X Visual acuity X X X X X Supplementation X X X Measurement of Xanthophylls Eye: MPOD (HRA) X X X X X Food frequency questionnaire X X Blood collection For (Heparin) Plasma to quantify Xanthophylls and Lipids X X X X X

Probands resident within a perimeter of 40km around the clinic will be preferentially selected to lower travel expenses. Recruitment takles place during regular visits in the course of the MACTEL study. For the angiography a vein will be punctated so that no additional punction is needed. Serum ist centrifuged at 1500g for 15min and kept at -70°C until analyse. Analyse of the Xanthophylls and Lipids in serum will be performed at the central laboratory of the University of Münster.

Autofluorescence imaging is part of study protocol for MACTEL Study. Two main images will be taken, one with an excitation wavelength of 488nm (good absorption by MP) and one with 514nm (poor absorption by MP). The digital subtration of both images provides a map of MP density around the fovea.

Inclusion criteria Informed consent Age at least 18y.? Type 2 IMT? Healthy general condition? At least one eye free from lens- or retina problems interfering with MP measurement with the modofied Heidelberg retina angiograph? Exclusion criteria No informed consent ? Younger than als 18 y.? Intake of Supplements containing L and Z (> 3mg L und >1mg Z) during the last 6 months? Bad general condition/ unintended loss of weight (>10%) within the last 3 monhs?

ELIGIBILITY:
Inclusion Criteria:

* Different distribution of macular pigment in patients with known macular teleangiectasia

Exclusion Criteria:

* No

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 12 patients with Macular Teleangiectasia
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2007-12; Study Completion 2008-02 (Estimated)

PRIMARY OUTCOMES:
Macular Pigment Optical Density | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Pauleikhoff, MD, Principal Investigator — Chairman Dep. of Ophthalmology, St.Franziskus Hospital, Muenster, Germany
Locations (1):
- Dep. of Ophthalmology, St. Franziskus Hospital, Münster, Germany